CLINICAL TRIAL: NCT05492097
Title: The Effect of Robot-assisted Walking Training on Balance, Trunk Control, Mobility, Spasticity and Motor Function in Hemiplegic Individuals
Brief Title: The Effect of Robot-assisted Walking Training on Hemiplegic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Principal Investigator, Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-667
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Hemiplegia; Gait, Hemiplegic; Motor Function; Balance; Distorted
MeSH Terms: conditions — Hemiplegia; Gait Disorders, Neurologic | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): For the patients in this group, 3 days a week for 4 weeks; various exercises and walking training will be given in sitting, crawling, kneeling, half-kneeling and standing positions and 20 minutes NMES will be applied.
  Interventions: Behavioral: Exercise Therapy
- Exercise and Robotic Group (Experimental): In addition to the exercise group treatment, patients will receive gait training for 4 weeks, 3 sessions a week, with the last effector fixed robot Lokohelp.
  Interventions: Behavioral: Exercise Therapy and Robotic Walking Training

INTERVENTIONS:
Behavioral: Exercise Therapy — Traditional exercise therapy and NMES
  Arms: Exercise Group
Behavioral: Exercise Therapy and Robotic Walking Training — Traditional exercise therapy and Robotic Walking Training
  Arms: Exercise and Robotic Group

SUMMARY:
The aim of this study is to compare the effects of robotic rehabilitation on balance, body control, mobility, spasticity, motor function and depression compared to traditional therapy in individuals with chronic stroke. Patients aged between 40-70 years, who applied to the Private Avrasya Hospital Physical Therapy and Rehabilitation Clinic, were diagnosed with hemiplegia based on an epicrisis medical board report, were included in the study on a voluntary basis, regardless of gender. After recording the demographic and clinical information of the participants, based on the physician's decision, they were included in 2 groups: conventional treatment combined with robotic rehabilitation (n=20) and conventional treatment only (n=20).

While one of the groups received traditional treatment, the other group received robotic walking training in addition to conventional treatment. Traditional treatment includes strengthening, balance, range of motion exercises and gait training applied 3 days a week for 4 weeks. Robot-assisted walking training was planned for 20 minutes, 3 days a week.

As assessment methods, number of steps, the 10m Walk Test, Brunnstrom motor staging, Functional Ambulation Classification, Fugl Meyer Rating Scale (lower extremity section), Modified Ashworth Scale, Beck Depression Scale, Tinetti Balance and Gait Test, Postural Assessment Scale in Stroke Patients and Stroke Impact Scale were used. Gender, age and duration of illness showed homogeneous distribution between the groups.

DETAILED DESCRIPTION:
More than 80% of stroke survivors have impaired walking ability, but most regain their ability to walk. While 40% of them need help while walking, 60% of the group do not have the ability to move independently outside the home. Balance disorder is the most common problem after stroke. Decreased muscle strength and joint range of motion and impaired coordination and sensory organization mechanism prevent balance. 80% of individuals who have had a stroke for the first time have balance disorder in the subacute phase. As a result of restricted balance, postural control deteriorates, the risk of falling increases and mobility decreases.

Interventions to improve gait function should be intense, repetitive, and task-oriented. Intensive efforts of more than one physiotherapist are required in patients who do not have independent gait. Robot assisted walking devices; provides high-intensity, repetitive, task-specific therapy. It both reduces the workload of physiotherapists and improves gait quality, functional results (walking speed and capacity) and motor performance with multi-sensory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Having had a stroke once and associated hemiplegia,
* At least 1 year has passed since the stroke,
* Stage 3 and above in terms of lower extremity recovery level according to the Brunnstrom motor staging scale,
* Level 2 and above according to the Functional Ambulation Classification

Exclusion Criteria:

* Concomitant peripheral nerve lesion or lower motor neuron disease;
* Presence of other neurological disorders such as ataxia, dyskinesia, dystonia;
* Any circulatory disorder
* Presence of advanced osteoporosis, arrhythmia, or serious heart condition;
* Advanced spasticity, peripheral lesion, pressure sore, advanced muscle atrophy, obesity, skin irritation, presence of cardiac pacemaker;
* Surgery or botulinum toxin administration in the last 6 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
The 10-meter walking test | 0-4 weeks
  The 10-meter walking test will be performed in the 16-meter walking area without looking at the first and last 3 meters. The stopwatch will be started after the patient walks for the first 3 meters and the time will be stopped after the 10 meters are completed. The time to complete the 10 meters will be determined in seconds.
Number of Steps | 0-4 weeks
  Calculation of the number of steps in one minute.
The Fugl Meyer Rating Scale | 0-4 weeks
  The Fugl Meyer Rating Scale is a scale used to evaluate sensorimotor impairment in individuals with stroke. The maximum score is 226, which corresponds to full sensory-motor recovery. It is an ordinal scale with 3 points for each item. A given task is given 0 points if it cannot be done, 1 point if it is partially done, and 2 points if it is done completely. Reflex activity is measured using only 2 points, 0 points are given if there is no reflex, and 2 points are given if there is. In the study, the 34-point part of the scale for the lower extremity will used.
The Postural Rating Scale in Stroke Patients | 0-4 weeks
  The Postural Rating Scale for Stroke Patients (PASS-Turk) will be used to assess trunk control. This scale helps to predict prognosis, shape treatment, and monitor time-dependent improvement. It is advantageous in that it is comprehensive, sensitive in evaluating changes in patients, and can be used even in patients with low physical capacity. The scale consists of 12 questions and each question is scored between 0-3 (0 = unable to do, 3 = able to do without assistance).
Tineti Balance and Gait Assessment | 0-4 weeks
  The scale consists of 2 subtests: the first 9 questions are about balance and the next 7 questions are about walking. In 16 questions, the movements during ADL are questioned. If the movement is done correctly, 2 points are given, if the movement is made with adaptations, 1 point is given, if it cannot be done, 0 points are given. If the total score is 18 and below, the risk of falling is high, if it is 19-24, the risk of falling is moderate, and if it is 24 and above, the risk of falling is high.
The Stroke Impact Scale | 0-4 weeks
  The Stroke Impact Scale will be used as a stroke-specific health status measure in the assessment of quality of life. It consists of a total of 59 items and 8 subsections: strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, participation. If the patient cannot complete the item, he will be asked to give 1 point, if he has no difficulty in completing it, he will be asked to give 5 points. At the end of the scale, the visual analog scale (0: No recovery, 100: Complete recovery) will evaluate the perception of general recovery after stroke.
Brunnstrom motor staging | 0-4 weeks
  Brunnstrom motor staging is a test that measures motor progress in parts of the central nervous system that regulate motor performance in patients with hemiplegia. The degree of recovery of the central nervous system is evaluated by enabling the patient to perform selected motor actions that require progressively better neuromuscular control. There are 6 stages for the lower extremity
Functional Ambulation Scale | 0-4 weeks
  The amount of physical support that patients need during walking will be determined by the Functional Ambulation Scale. Evaluation is made out of 6 points between 0-5 (0=Cannot ambulatory alone, 5=Can walk independently on all kinds of surfaces).
The Modified Ashworth Scale | 0-4 weeks
  The Modified Ashworth Scale is the most commonly used assessment method for spasticity in the international arena (10). The patient is examined in a supine and relaxed position. The joint is moved passively, repetitively and rapidly, and is scored between 0 and 4 according to the resistance of the joint to movement (0 = no increase in tone, 4 = the affected extremity is rigid in flexion and extension).
Beck Depression Scale | 0-4 weeks
  Emotional symptoms such as hopelessness and guilt and physical symptoms such as weight loss, fatigue and insomnia are also examined in the questions in the scale. There are 21 questions, points are given between 0-3. According to the total score, it is evaluated as follows: 0 to 9 points = minimal depressive symptoms, 10 to 16 points = mild depressive symptoms, 17 to 29 points = moderate depressive symptoms, 30 to 63 points = severe depressive symptoms .

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)